CLINICAL TRIAL: NCT01709240
Title: Evaluation of the BioWeld1 System as a Method for Surgical Incision Closure
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Internal decision
Sponsor: IonMed Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BW102
Record Dates: First submitted 2012-10-16; First posted 2012-10-18 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2012-10

CONDITIONS: Child Delivery Using an Elective C- Section
Keywords: Chitosan; Plasma; Incision Closure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BioWeld1 System (Experimental)
  Interventions: Device: BioWeld1 System

INTERVENTIONS:
Device: BioWeld1 System — External skin layer closure of C-section incision by the BioWeld1 system. Removal of Chitoplast on day 4-7 post procedure.

SUMMARY:
The purpose of this study is to assess the safety and performance of the BioWeld1 System procedure for surgical incision closure of the skin in women scheduled for elective C-section procedure.

DETAILED DESCRIPTION:
In every surgical procedure, there is a need to close the incision that was made. Current methods for incision closure include stitching, gluing and stapling. Some of these methods are time consuming, have potential for infection and may leave a significant scar. The bioWeld1 technology suggests a new approach for incision closure. It is a novel medical device that consists of a Chitosan film and the BioWeld1 plasma ejecting device. The Chitosan film is intended to be applied to the skin incision, while the BioWeld1device is used for welding the Chitosan to the skin by means of cold plasma technology.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 to 40 years old.
2. Women scheduled for child delivery using an elective C- section.
3. Women in their first or second pregnancy having a C-section for the first time
4. Healthy women with no systemic diseases such as diabetes, heart disease etc.
5. Women with average weight, BMI prior pregnancy of 18.5-25.
6. Women with no skin diseases
7. Subject understands the study requirements and the treatment procedures and provides written Informed Consent before any study-specific tests or procedures are performed.
8. The subject commits to return for the scheduled post-operative follow-up visits at the clinic

General Exclusion Criteria:

1. Women intended for any abdominal surgery other than C-section procedure
2. Women intended for C-section procedure for other purpose than child delivery
3. Any prior C-section procedure for any purpose
4. Women Received/Receiving radiotherapy or chemotherapy of any kind.
5. Women receiving steroids or any other medication that interferes with wound healing.
6. Women receiving Acutan in the last half year.
7. Women with bleeding diathesis or hypercoagulable state.
8. Women with prior cosmetic or medical treatment in the target area (e.g. phosphatydilcholine injections).
9. Women suffering from Thrombocytopenia (platelets count<100,000/mm3) pre-procedure.
10. Women who is currently participating or have participated in an investigational study, other than this study, within the past 60 days.
11. Psychiatric background.

Intra operative exclusion criteria:

1. Severe excessive bleeding from the wound
2. Patient is not eligible for an experimental closure according to the physician discretion.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2013-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Safety | Within 21 days post procedure
  Frequency and severity of incision closure procedure-related adverse events (burns, wound dehiscence or need for additional surgical procedure of the skin wound).

SECONDARY OUTCOMES:
Performance | At 21 days post procedure
  The following secondary variables will be examined:
  1. Complete epidermal closure.
  2. Redness and edemas grade <1 in at least 87% of the subjects.
  3. Encrustation grade <1 in at least 87% of the subjects.
  4. Discharge from wound is negative in at least 87% of the subjects.
  5. Photographic evidence of clean healing in at least 30% of the cases.

CONTACTS AND LOCATIONS:
Overall Officials: Drorit Hochner-Celnikier, MD, Principal Investigator — Hadassah University Hospital, Mount Scopus
Locations (1):
- Hadassah University Hospital, Mount Scopus, Jerusalem, Israel, Israel